CLINICAL TRIAL: NCT01766973
Title: Observational Study to Determine Abnormalities in Resting State fMRI in Chronic Back Pain.
Brief Title: Decoding Chronic Pain With fMRI
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr Ben Seymour, Wellcome Intermediate Clinical Fellow, University of Cambridge
Other Study IDs: CE-U.NA.NFLT.EGDF
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Chronic Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic back pain: Adults, >6months duration
- Control: Age and sex matched controls

SUMMARY:
Recent evidence suggests that chronic pain is associated with abnormal connectivity between brain regions associated with the processing of pain. We aim to test the diagnostic power of resting state functional magnetic resonance imaging (MRI) to diagnose patients with chronic back pain. Using new methods of image acquisition and analysis we aim to develop a computational method to correctly classify patients and matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60
* pain > 6months
* right-handed
* non-smoking
* mechanical back pain

Exclusion Criteria:

* significant neurological or psychiatric disease
* major systemic illness
* MRI exclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults with >6 months of mechanical lower back pain, not sue to any major systemic disease
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-04-06 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Functional brain connectivity | 6 months
  Assessed by fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Ben Seymour, MRCP PhD, Principal Investigator — University of Cambridge
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom